CLINICAL TRIAL: NCT05831813
Title: The Feasibility, Acceptability and Preliminary Efficacy of a Group Intervention Aimed at Reducing Social and Emotional Loneliness: a Pilot Study
Brief Title: The Feasibility, Acceptability and Preliminary Efficacy of a Group Intervention to Reduce Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Responsible Party: Principal Investigator, Carmen van den Bulck, C.M.M. (Carmen) van den Bulck, MSc, University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-CP-15875
Record Dates: First submitted 2023-02-14; First posted 2023-04-26 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Loneliness; Social Isolation
Keywords: Loneliness; Social Isolation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: Before the intervention starts, participants will first follow a baseline period, ranging between 1 and 7 weeks. The length of the baseline period is based on the date of enrolment and therefore not random. Following the baseline period, all participants will start in the group intervention. Data are collected at screening, pre-intervention, post-intervention, one-month follow-up and three-month follow-up, as well as during weekly measurements during the waiting list period and the course.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Goal-Based Cognitive Behavioural Intervention (Experimental): Participants start with a 1 to 7 weeks baseline period. The duration is based on the enrolment date and therefore not random. Afterward, all participants enter the intervention, which promotes social behavioural activation aligned with personal values and teaches skills that make negative emotions and thoughts less bothersome and reduce feelings of loneliness. The intervention comprises seven weekly sessions and a follow-up, conducted in a group format to facilitate interpersonal practice and is presented as a course for enhanced acceptability.
  Please note: The original design involved an RCT with a Goal-Based Cognitive Behavioral Intervention as the experimental arm and a waitlist arm. Participants in the waitlist arm would enter the intervention after a waitlist period. Due to limited enrollments, the design was modified to a single arm resembling the waitlist arm of the initial RCT design.
  Interventions: Behavioral: Goal-Based Cognitive Behavioural Intervention

INTERVENTIONS:
Behavioral: Goal-Based Cognitive Behavioural Intervention — A goal-based cognitive behavioural intervention in a group format that addresses negative social cognitions and focuses on social approach processes

SUMMARY:
Severe loneliness is a large and growing clinical and societal problem. Although there are interventions for loneliness, elevated levels often remain. This pilot study evaluates the feasibility and acceptability of an intervention to alleviate social and emotional loneliness among students. The second aim is to obtain effect sizes that inform sample size calculations of a subsequent randomized controlled trial (RCT). The goal of this clinical trial is to learn about the feasibility and acceptability of a group intervention aimed at reducing social and emotional loneliness and social isolation in students. In addition, we want to obtain effect sizes that can inform the sample size calculation of a subsequent randomized controlled trial (RCT).

The hypotheses are that:

* Participants after completing the intervention have reduced levels of social and emotional loneliness and social isolation compared to baseline (primary outcomes).
* Participants after completing the intervention have reduced levels of social anxiety, depressive symptoms, and better daily functioning compared to baseline (secondary outcomes).

Before the group intervention starts, participants will first follow a baseline period, ranging between 1 and 7 weeks. The length of the baseline period is based on the date of enrolment and therefore not random. Following the baseline period, all participants will start in the group intervention. This intervention aims to encourage social behavioural activation tailored to the values of the participant and teach skills that make negative emotions and thoughts less bothersome and reduce feelings of loneliness. This intervention consists of seven weekly group sessions and a booster session. The intervention is offered in a group format to maximize possibilities for interpersonal therapeutic practice and is framed as a psycho-educational course to increase its acceptability.

Data are collected at screening, pre-intervention, post-intervention, one-month follow-up and three-month follow-up, as well as during weekly measurements during the baseline period and the course period. Primary outcome measures are social and emotional loneliness and social isolation. Secondary outcome measures are social anxiety, depression, and daily functioning. Other outcome measures are interpersonal problems and assessment of the sessions.

Participants will be recruited via posters at the University of Amsterdam.

ELIGIBILITY:
Inclusion criteria:

* Being at least 16 years old
* Exhibiting at least moderate levels of loneliness as assessed by the De Jong Gierveld Loneliness Scale 11-item version (DJGLS; de Jong-Gierveld & Kamphuls, 1985)
* Possessing sufficient proficiency in the English language.

Exclusion criteria:

- The presence of severe (psychiatric) problems that hinder participation in the study or require other forms of immediate care, as indicated by the Mini International Neuropsychiatric Interview 7.0.2 (MINI; Sheehan et al., 1998).

If participants were already receiving psychological or pharmacological treatment for psychiatric problems, this treatment had to be temporarily interrupted for the duration of the study in consultation with the participant's clinician.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-11 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Changes in social loneliness | Assessed at screening (1 to 8 weeks before pretest), pretest, posttest (8 weeks after pretest), one-month follow-up and three-month follow-up.
  Loneliness Scale (LS; de Jong Gierveld & van Tilburg, 1999). The 11-item Loneliness Scale was used to measure emotional and social loneliness. Participants score the items on a 5-point Likert scale ("yes!", "yes", "more or less", "no", "no!").
Weekly changes in social loneliness | Assessed in weekly measurements in the baseline period (up to 7 weeks before pretest) and in weekly measurements in the intervention period (up to 7 weeks after pretest)
  Loneliness Scale (LS; de Jong Gierveld & van Tilburg, 2006) The 6-item Loneliness Scale was used to measure emotional and social loneliness. Participants score the items on a 5-point Likert scale ("yes!", "yes", "more or less", "no", "no!").
Changes in emotional loneliness | Assessed at screening (1 to 8 weeks before pretest), pretest, posttest (8 weeks after pretest), one-month follow-up and three-month follow-up.
  Measured by the Loneliness Scale (LS; de Jong Gierveld & van Tilburg, 1999). The 11-item Loneliness Scale was used to measure emotional and social loneliness. Participants score the items on a 5-point Likert scale ("yes!", "yes", "more or less", "no", "no!").
Weekly changes in emotional loneliness | Assessed in weekly measurements in the baseline period (up to 7 weeks before pretest) and in weekly measurements in the intervention period (up to 7 weeks after pretest)
  Loneliness Scale (LS; de Jong Gierveld & van Tilburg, 2006) The 6-item Loneliness Scale was used to measure emotional and social loneliness. Participants score the items on a 5-point Likert scale ("yes!", "yes", "more or less", "no", "no!").
Changes in social isolation | Assessed at screening (1 to 8 weeks before pretest), pretest, posttest (8 weeks after pretest), one-month follow-up and three-month follow-up.
  Lubben Social Network Scale (LSNS; Lubben, 1998). The 12-item LSNS-R quantifies social isolation from family and friends. Participants score the items on a 6-point Likert scale.
Weekly changes in social isolation | Assessed in weekly measurements in the baseline period (up to 7 weeks before pretest) and in weekly measurements in the intervention period (up to 7 weeks after pretest)
  Lubben Social Network Scale (LSNS; Lubben, 2006). The 6-item LSNS quantifies social isolation from family and friends. Participants score the items on a 6-point Likert scale (0 ≥ 9 relatives/friends to 5 = no relatives/friends).

SECONDARY OUTCOMES:
Changes in depressive symptoms | Assessed at screening (1 to 8 weeks before pretest), pretest, posttest (8 weeks after pretest), one-month follow-up and three-month follow-up.
  Center for Epidemiological Studies Depression Scale (CES-D; Radloff, 1977). The 20-item CES-D was used to measure feelings of depression. Participants score the items on a 4-point scale, from "Rarely or none of the time (Less than 1 Day)" to "Most or all of the time (5-7 days)".
Changes in social anxiety | Assessed at screening (1 to 8 weeks before pretest), pretest, posttest (8 weeks after pretest), one-month follow-up and three-month follow-up.
  Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998). The SIAS is a 20-item questionnaire to assess social anxiety symptoms, specifically from the perspective of the individual when engaging in social interactions. Items are rated on a 5-point Likert scale (0 = not at all, 4 = very much).
Changes in daytime functioning | Assessed at screening (1 to 8 weeks before pretest), pretest, posttest (8 weeks after pretest), one-month and three-month follow-up, in weekly measurements in baseline period and intervention period (up to 7 weeks before and after pretest respectively)
  Daytime functioning (Hawkley et al.,2010) To measure daily functioning, the questionnaire 5-item questionnaire from Hawkley et al. (2010) rates the extent of sleepiness, exhaustion, liveliness, energy, and fatigue over the last seven days on a 5-point scale ("Not at all" to "Very much").

OTHER OUTCOMES:
Satisfaction of the followed sessions | Assessed in the seven weekly measurements in the intervention period (up to 7 weeks after pretest)
  Session Rating Scale 3.0 (SRS 3.0; Duncan et al., 2003) The SRS 3.0 is a 4-item visual analogue scale to assess the working alliance with the trainer and includes gathering information about how the client feels about the relationship with the trainer, the goals and topics of the session, the approach or method used, and an overall rating of the session.
Problematic interpersonal styles | Assessed at screening (1 to 8 weeks before pretest), pretest, posttest (8 weeks after pretest), one-month follow-up and three-month follow-up.
  Inventory of Interpersonal Problems-32 (IIP-32; Barkham et al.,1996). The 32-item IIP-32 was used to measure problematic interpersonal styles and consists of eight subscales (Domineering/ Controlling, Self-Serving/ Vindictive, Cold/ Distant, Avoidant/ Socially Inhibited, Non-assertive/ Obsequious, Exploitable/ Overly Accommodating, Overly Nurturant/ Self-Sacrificing, Intrusive/ Needy). The items are rated on a 5-point scale ("Not at all" to "Extremely").

CONTACTS AND LOCATIONS:
Overall Officials: Carmen van den Bulck, MSc, Principal Investigator — University of Amsterdam
Locations (1):
- University of Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Anonymised individual participant data underlying the results reported in this article will be available upon request.

REFERENCES:
- [Background] Alden LE, Buhr K, Robichaud M, Trew JL, Plasencia ML. Treatment of social approach processes in adults with social anxiety disorder. J Consult Clin Psychol. 2018 Jun;86(6):505-517. doi: 10.1037/ccp0000306. PMID 29781649
- [Background] Alden LE, Taylor CT. Relational treatment strategies increase social approach behaviors in patients with Generalized Social Anxiety Disorder. J Anxiety Disord. 2011 Apr;25(3):309-18. doi: 10.1016/j.janxdis.2010.10.003. Epub 2010 Oct 20. PMID 21094019
- [Background] Cacioppo S, Grippo AJ, London S, Goossens L, Cacioppo JT. Loneliness: clinical import and interventions. Perspect Psychol Sci. 2015 Mar;10(2):238-49. doi: 10.1177/1745691615570616. PMID 25866548
- [Background] Cacioppo JT, Hawkley LC. Perceived social isolation and cognition. Trends Cogn Sci. 2009 Oct;13(10):447-54. doi: 10.1016/j.tics.2009.06.005. Epub 2009 Aug 31. PMID 19726219
- [Background] Masi CM, Chen HY, Hawkley LC, Cacioppo JT. A meta-analysis of interventions to reduce loneliness. Pers Soc Psychol Rev. 2011 Aug;15(3):219-66. doi: 10.1177/1088868310377394. Epub 2010 Aug 17. PMID 20716644
- [Background] Qualter P, Vanhalst J, Harris R, Van Roekel E, Lodder G, Bangee M, Maes M, Verhagen M. Loneliness across the life span. Perspect Psychol Sci. 2015 Mar;10(2):250-64. doi: 10.1177/1745691615568999. PMID 25910393

DOCUMENTS (1):
  • Informed Consent Form (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT05831813/ICF_000.pdf